CLINICAL TRIAL: NCT01887158
Title: Phase 4 Study of Comparison of 2-Liter Mixed Preparation With Bisacodyl Plus Polyethylene Glycol and 4-Liter Polyethylene Glycol for Colon Cleansing in Patients With Prior History of Colorectal Resection. A Prospective Randomized Controlled Trial.
Brief Title: Efficacy of 2-Liter Mixed Preparation With Bisacodyl Plus Polyethylene Glycol and 4-Liter Polyethylene Glycol for Colon Cleansing in Patients With Prior History of Colorectal Resection
Acronym: PEGOP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ospedale Santa Maria delle Croci (Other)
Responsible Party: Principal Investigator, Alessandro Mussetto, MD, Ospedale Santa Maria delle Croci
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PEGOP0613
Record Dates: First submitted 2013-06-11; First posted 2013-06-26 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-06

CONDITIONS: Intestinal Cancer
MeSH Terms: conditions — Intestinal Neoplasms | interventions — Polyethylene Glycols; Bisacodyl

STUDY DESIGN:
Who Masked: Care Provider

ARMS (2):
- bisacodyl plus 2-Liter Polyethylene glycol (Active Comparator): Patients randomized to the low-volume arm, will be invited to consume 2 sachets of Lovol-esse (Polyethylene glycol) in one liter of water at 8:00 PM the evening before the colonoscopy and 2 sachets in one liter of water 4 hours before their scheduled colonoscopy appointment; furthermore, the patients will be instructed to take three 5-mg tablets of bisacodyl the day before the procedure, at 5:00 PM.
  Interventions: Drug: Polyethylene glycol; Drug: Bisacodyl
- 4-Liter Polyethylene glycol (Active Comparator): Patients assigned to the high-volume arm will be invited to consume 2 envelopes of Selg-esse 1000 (polyethylene glycol) in 2 litres of water and drink the resulting solution in about 2-3 hours starting at 6:00 PM the evening before the colonoscopy; the day of the procedure, starting 5 hours before the procedure, the patients will be invited to complete the preparation with 2 others envelopes of Selg-esse 1000 (polyethylene glycol) dissolved in 2 litres of water.
  Interventions: Drug: Polyethylene glycol

INTERVENTIONS:
Drug: Polyethylene glycol
Drug: Bisacodyl
  Arms: bisacodyl plus 2-Liter Polyethylene glycol

SUMMARY:
Studies that have investigated different bowel preparations in patients with history of colorectal surgery are surprisingly lacking.Therefore, which is the best colon preparation in this subgroup of patients is still unknown. Polyethylene glycol (PEG)-based solutions are the most popular and safest bowel preparation regimens, however the 4-Liter volume is often poorly tolerated. More recently, it has been shown that the use of a low volume preparation (2-Liter PEG solution with the adjunct of a laxative, bisacodyl) achieves comparable bowel cleanliness rates to 4-Liter PEG in general population.The primary aim will be to compare the efficacy of 2-L mixed preparation (bisacodyl plus PEG) to 4-L PEG preparation.

ELIGIBILITY:
Inclusion Criteria:

1. Outpatients
2. ≥18 yrs old,
3. Prior history of colorectal resection due to colo-rectal cancer, referred for surveillance colonoscopy

Exclusion Criteria:

1. Inpatients
2. Emergency Colonoscopy
3. Comorbidities: Congestive heart failure, history of kidney disease, history of solid organ transplant
4. Pregnant and/or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2013-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
quality of bowel preparation rated according to a modified Ottawa bowel preparation scale | about 2 weeks after the randomization

SECONDARY OUTCOMES:
Tolerability to the preparation (specific questionaire) | participants will be followed from the randomization until the time of colonoscopy, about 2 weeks after the randomization
  Tolerability will be assessed by using a questionnaire completed by the patients on arrival at the endoscopy unit before colonoscopy.
  The patient acceptance/satisfaction to bowel preparation will be evaluated with the following question:
  What is the extent of your disturbance due to bowel preparation? Severe (the bowel preparation assumption was stopped and not completed)(score 3) Moderate (bowel preparation assumption was stopped several times because of side effects but finally completed)(score 2) Mild (bowel preparation was completed without pauses but with some mild side effects)(score 1) No side effects (score 0)
safety (adverse event rate) | participants will be followed from the randomization until the time of colonoscopy, about 2 weeks after the randomization
  Safety will be evaluated through reported adverse events, physical examination and vital signs
Lesion detection (type and lesion detection rate/patient) | about 2 weeks from the randomization
  Polyps will be categorized as non-neoplastic or neoplastic (ie, adenomatous). Adenoma will be diagnosed by pathological evaluation of retrieved polyps. Adenomas will be considered advanced when they will be ≥10 mm in size, with villous architecture, high-grade dysplasia or intramucosal carcinoma (pTis), or 3 or more adenomas will be found. Invasive cancer will be considered when malignant cells will be observed beyond the muscularis mucosa. Size of adenoma will be obtained from both the colonoscopist's assessment and the pathology report, with the larger measurement being used in the analyses. Site of adenoma will be recorded by the colonoscopist at the time of polypectomy. Lesions at or proximal to the splenic flexure will be termed right-sided lesions, those distal to the splenic flexure as left-sided, taking into account the type of colorectal surgical resection underwent by the patient. The adenoma detection rate will be defined as the proportion of colonoscopies with adenomas.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Alessandro Mussetto, Ravenna, RA
  - Ospedale S.Maria delle Croci, Ravenna, RA

REFERENCES:
- [Derived] Mussetto A, Frazzoni L, Paggi S, Dari S, Laterza L, Radaelli F, Hassan C, Triossi O, Fuccio L. Split dosing with a low-volume preparation is not inferior to split dosing with a high-volume preparation for bowel cleansing in patients with a history of colorectal resection: a randomized trial. Endoscopy. 2015 Oct;47(10):917-24. doi: 10.1055/s-0034-1391987. Epub 2015 Apr 24. PMID 25910064